CLINICAL TRIAL: NCT07381192
Title: An Artificial Intelligence System for Multimodal, Multi-class Diagnosing Solid Pancreatic Lesions Based on Endoscopic Ultrasound
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Liaocheng People's Hospital (Other); Taian City Central Hospital (Other); Qilu Hospital of Shandong University (Qingdao) (Other); Binzhou People's Hospital (Other); Shandong Provincial Hospital (Other Government); The Affiliated Hospital of Qingdao University (Other); Qianfoshan Hospital (Other); Shengli Oilfield Hospital (Other); Binzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: 2025-SDU-QILU-6
Record Dates: First submitted 2025-12-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-09

CONDITIONS: Endoscopic Ultrasound (EUS); Solid Pancreatic Lesion
Keywords: endoscopic ultrasound; solid pancreatic lesion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Endoscopic ultrasound images, endoscopic ultrasound features, clinical data and imaging features from patients who underwent endoscopic ultrasound.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing EUS: Patients aged ≥18 years scheduled for EUS with suspected solid pancreatic lesions based on clinical symptoms, medical history, laboratory tests or radiological examinations agree to participate in the research and be able to sign informed consent.
  Interventions: Device: iEUS-SPL(intelligent endoscopic ultrasound system-pancreatic solid lesion)

INTERVENTIONS:
Device: iEUS-SPL(intelligent endoscopic ultrasound system-pancreatic solid lesion) — The iEUS-SPL will automaticly detect solid pancreatic lesions and integrate the patients' endoscopic ultrasound images, endoscopic ultrasound features, clinical data and imaging features to perform a five-category classification for the lesions, categorizing them as pancreatic cancer, pancreatic neuroendocrine tumor, solid pseudopapillary tumor, autoimmune pancreatitis and chronic pancreatitis.

SUMMARY:
The aim of this study is to validate an artificial intelligence system named iEUS-SPL(intelligent endoscopic ultrasound system-solid pancreatic lesion) for detecting and multimodal, multi-class diagnosing solid pancreatic lesions during endoscopic ultrasound(EUS) examination.

DETAILED DESCRIPTION:
This is an observational study with a prospective, cohort design. We have developed an artificial intelligence system named iEUS-SPL for multimodal, multi-class diagnosing solid pancreatic lesions using endoscopic ultrasound images, endoscopic ultrasound features, clinical data and imaging features from retrospectively collected patients who underwent EUS. The lesion detection rate and diagnostic performance of iEUS-SPL in identifying solid pancreatic lesions will be evaluated in real-time EUS scanning videos over prospective enrolled cases.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥18 years scheduled for EUS with suspected solid pancreatic lesions based on clinical symptoms, medical history, laboratory tests or radiological examinations agree to participate in the research and be able to sign informed consent.
2. Patients with no prior history of treatment for pancreatic lesions.

Exclusion Criteria:

1. Patients with absolute contraindications to EUS examination.
2. Pregnancy or lactating.
3. Uncorrectable coagulopathy(PTT>50 seconds or INR>1.5) and/or uncorrectable thrombocytopenia(platelet count<50×109/L).
4. Upper gastrointestinal obstruction.
5. Patients who underwent surgical treatment or anatomical alterations of the pancreas due to lesions in other thoracic and/or abdominal organs, as well as patients with congenital anatomical abnormalities.
6. Patients who have undergone biliary/pancreatic duct stent placement.
7. Patients who refuse to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with suspected solid pancreatic lesions undergoing EUS.
Sampling Method: Non-Probability Sample
Enrollment: 383 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
The accuracy of iEUS-SPL for solid pancreatic lesions | During procedure
  The primary outcome of the study is to evaluate the accuracy of the iEUS-SPL in identifying the solid pancreatic lesions (including pancreatic cancer, pancreatic neuroendocrine tumor, solid pseudopapillary tumor, autoimmune pancreatitis, chronic pancreatitis).
The sensitivity of iEUS-SPL for solid pancreatic lesions | During procedure
  The primary outcome of the study is to evaluate the sensitivity of the iEUS-SPL in identifying the solid pancreatic lesions (including pancreatic cancer, pancreatic neuroendocrine tumor, solid pseudopapillary tumor, autoimmune pancreatitis, chronic pancreatitis).
The specificicy of iEUS-SPL for solid pancreatic lesions | During procedure
  The primary outcome of the study is to evaluate the specificity of the iEUS-SPL in identifying the solid pancreatic lesions (including pancreatic cancer, pancreatic neuroendocrine tumor, solid pseudopapillary tumor, autoimmune pancreatitis, chronic pancreatitis).
The postive predictive value of iEUS-SPL for solid pancreatic lesions | During procedure
  The primary outcome of the study is to evaluate the postive predictive value of the iEUS-SPL in identifying the solid pancreatic lesions (including pancreatic cancer, pancreatic neuroendocrine tumor, solid pseudopapillary tumor, autoimmune pancreatitis, chronic pancreatitis).
The negative predictive value of iEUS-SPL for solid pancreatic lesions | During procedure
  The primary outcome of the study is to evaluate the negative predictive value of the iEUS-SPL in identifying the solid pancreatic lesions (including pancreatic cancer, pancreatic neuroendocrine tumor, solid pseudopapillary tumor, autoimmune pancreatitis, chronic pancreatitis).
the lesion detection rate of iEUS-SPL for detecting solid pancreatic lesions | During procedure
  The primary outcome of the study is to evaluate the lesion detection rate of the iEUS-SPL in identifying the solid pancreatic lesions(defined as the number of detected lesions divided by the total number of lesions).

SECONDARY OUTCOMES:
Comparison of the accuracy between iEUS-SPL and endosonographers | During procedure
  The secondary outcome of the study is to comparing the accuracy between iEUS-SPL and different-level endosonographers in identifying the solid pancreatic lesions (including pancreatic cancer, pancreatic neuroendocrine tumor, solid pseudopapillary tumor, autoimmune pancreatitis, chronic pancreatitis).
Comparison of the sensitivity between iEUS-SPL and endosonographers | During procedure
  The secondary outcome of the study is to comparing the sensitivity between iEUS-SPL and different-level endosonographers in identifying the solid pancreatic lesions (including pancreatic cancer, pancreatic neuroendocrine tumor, solid pseudopapillary tumor, autoimmune pancreatitis, chronic pancreatitis).
Comparison of the specificity between iEUS-SPL and endosonographers | During procedure
  The secondary outcome of the study is to comparing the specificity between iEUS-SPL and different-level endosonographers in identifying the solid pancreatic lesions (including pancreatic cancer, pancreatic neuroendocrine tumor, solid pseudopapillary tumor, autoimmune pancreatitis, chronic pancreatitis).
Comparison of the postive predictive value between iEUS-SPL and endosonographers | During procedure
  The secondary outcome of the study is to comparing the postive predictive value between iEUS-SPL and different-level endosonographers in identifying the solid pancreatic lesions (including pancreatic cancer, pancreatic neuroendocrine tumor, solid pseudopapillary tumor, autoimmune pancreatitis, chronic pancreatitis).
Comparison of the negative predictive value between iEUS-SPL and endosonographers | During procedure
  The secondary outcome of the study is to comparing the negative predictive value between iEUS-SPL and different-level endosonographers in identifying the solid pancreatic lesions (including pancreatic cancer, pancreatic neuroendocrine tumor, solid pseudopapillary tumor, autoimmune pancreatitis, chronic pancreatitis).

CONTACTS AND LOCATIONS:
Locations (1):
- Qilu Hospital of Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bang JY, Saftoiu A, Udristoiu A, Gruionu L, Codruta Gheorghe E, Gruionu G, Ramesh J, Wilcox CM, Varadarajulu S. Prospective clinical validation of a novel artificial intelligence system for real-time detection of solid pancreatic masses during endoscopic ultrasonography. Endoscopy. 2025 Oct 13. doi: 10.1055/a-2701-6530. Online ahead of print. PMID 40953587
- [Background] Cui H, Zhao Y, Xiong S, Feng Y, Li P, Lv Y, Chen Q, Wang R, Xie P, Luo Z, Cheng S, Wang W, Li X, Xiong D, Cao X, Bai S, Yang A, Cheng B. Diagnosing Solid Lesions in the Pancreas With Multimodal Artificial Intelligence: A Randomized Crossover Trial. JAMA Netw Open. 2024 Jul 1;7(7):e2422454. doi: 10.1001/jamanetworkopen.2024.22454. PMID 39028670
- [Background] Wu HL, Yao LW, Shi HY, Wu LL, Li X, Zhang CX, Chen BR, Zhang J, Tan W, Cui N, Zhou W, Zhang JX, Xiao B, Gong RR, Ding Z, Yu HG. Validation of a real-time biliopancreatic endoscopic ultrasonography analytical device in China: a prospective, single-centre, randomised, controlled trial. Lancet Digit Health. 2023 Nov;5(11):e812-e820. doi: 10.1016/S2589-7500(23)00160-7. Epub 2023 Sep 27. PMID 37775472
- [Background] Zhang J, Zhu L, Yao L, Ding X, Chen D, Wu H, Lu Z, Zhou W, Zhang L, An P, Xu B, Tan W, Hu S, Cheng F, Yu H. Deep learning-based pancreas segmentation and station recognition system in EUS: development and validation of a useful training tool (with video). Gastrointest Endosc. 2020 Oct;92(4):874-885.e3. doi: 10.1016/j.gie.2020.04.071. Epub 2020 May 6. PMID 32387499
- [Background] Oh CK, Kim T, Cho YK, Cheung DY, Lee BI, Cho YS, Kim JI, Choi MG, Lee HH, Lee S. Convolutional neural network-based object detection model to identify gastrointestinal stromal tumors in endoscopic ultrasound images. J Gastroenterol Hepatol. 2021 Dec;36(12):3387-3394. doi: 10.1111/jgh.15653. Epub 2021 Aug 16. PMID 34369001
- [Background] Dahiya DS, Al-Haddad M, Chandan S, Gangwani MK, Aziz M, Mohan BP, Ramai D, Canakis A, Bapaye J, Sharma N. Artificial Intelligence in Endoscopic Ultrasound for Pancreatic Cancer: Where Are We Now and What Does the Future Entail? J Clin Med. 2022 Dec 16;11(24):7476. doi: 10.3390/jcm11247476. PMID 36556092
- [Background] Kim YH, Kim GH, Kim KB, Lee MW, Lee BE, Baek DH, Kim DH, Park JC. Application of A Convolutional Neural Network in The Diagnosis of Gastric Mesenchymal Tumors on Endoscopic Ultrasonography Images. J Clin Med. 2020 Sep 29;9(10):3162. doi: 10.3390/jcm9103162. PMID 33003602
- [Background] Qin X, Zhang M, Zhou C, Ran T, Pan Y, Deng Y, Xie X, Zhang Y, Gong T, Zhang B, Zhang L, Wang Y, Li Q, Wang D, Gao L, Zou D. A deep learning model using hyperspectral image for EUS-FNA cytology diagnosis in pancreatic ductal adenocarcinoma. Cancer Med. 2023 Aug;12(16):17005-17017. doi: 10.1002/cam4.6335. Epub 2023 Jul 17. PMID 37455599
- [Background] Tian S, Shi H, Chen W, Li S, Han C, Du F, Wang W, Wen H, Lei Y, Deng L, Tang J, Zhang J, Lin J, Shi L, Ning B, Zhao K, Miao J, Wang G, Hou H, Huang X, Kong W, Jin X, Ding Z, Lin R. Artificial intelligence-based diagnosis of standard endoscopic ultrasonography scanning sites in the biliopancreatic system: a multicenter retrospective study. Int J Surg. 2024 Mar 1;110(3):1637-1644. doi: 10.1097/JS9.0000000000000995. PMID 38079604
- [Background] Oh S, Kim YJ, Park YT, Kim KG. Automatic Pancreatic Cyst Lesion Segmentation on EUS Images Using a Deep-Learning Approach. Sensors (Basel). 2021 Dec 30;22(1):245. doi: 10.3390/s22010245. PMID 35009788
- [Background] Norton ID, Zheng Y, Wiersema MS, Greenleaf J, Clain JE, Dimagno EP. Neural network analysis of EUS images to differentiate between pancreatic malignancy and pancreatitis. Gastrointest Endosc. 2001 Nov;54(5):625-9. doi: 10.1067/mge.2001.118644. PMID 11677484
- [Background] Nakamura H, Fukuda M, Matsuda A, Makino N, Kimura H, Ohtaki Y, Nawa Y, Oyama S, Suzuki Y, Kobayashi T, Ishizawa T, Kakizaki Y, Ueno Y. Differentiating localized autoimmune pancreatitis and pancreatic ductal adenocarcinoma using endoscopic ultrasound images with deep learning. DEN Open. 2024 Mar 2;4(1):e344. doi: 10.1002/deo2.344. eCollection 2024 Apr. PMID 38434146
- [Background] Dhali A, Kipkorir V, Srichawla BS, Kumar H, Rathna RB, Ongidi I, Chaudhry T, Morara G, Nurani K, Cheruto D, Biswas J, Chieng LR, Dhali GK. Artificial intelligence assisted endoscopic ultrasound for detection of pancreatic space-occupying lesion: a systematic review and meta-analysis. Int J Surg. 2023 Dec 1;109(12):4298-4308. doi: 10.1097/JS9.0000000000000717. PMID 37800594
- [Background] Das A, Nguyen CC, Li F, Li B. Digital image analysis of EUS images accurately differentiates pancreatic cancer from chronic pancreatitis and normal tissue. Gastrointest Endosc. 2008 May;67(6):861-7. doi: 10.1016/j.gie.2007.08.036. Epub 2008 Jan 7. PMID 18179797
- [Background] Kuwahara T, Hara K, Mizuno N, Haba S, Okuno N, Kuraishi Y, Fumihara D, Yanaidani T, Ishikawa S, Yasuda T, Yamada M, Onishi S, Yamada K, Tanaka T, Tajika M, Niwa Y, Yamaguchi R, Shimizu Y. Artificial intelligence using deep learning analysis of endoscopic ultrasonography images for the differential diagnosis of pancreatic masses. Endoscopy. 2023 Feb;55(2):140-149. doi: 10.1055/a-1873-7920. Epub 2022 Jun 10. PMID 35688454
- [Background] Tian G, Xu D, He Y, Chai W, Deng Z, Cheng C, Jin X, Wei G, Zhao Q, Jiang T. Deep learning for real-time auxiliary diagnosis of pancreatic cancer in endoscopic ultrasonography. Front Oncol. 2022 Oct 7;12:973652. doi: 10.3389/fonc.2022.973652. eCollection 2022. PMID 36276094
- [Background] Qin X, Ran T, Chen Y, Zhang Y, Wang D, Zhou C, Zou D. Artificial Intelligence in Endoscopic Ultrasonography-Guided Fine-Needle Aspiration/Biopsy (EUS-FNA/B) for Solid Pancreatic Lesions: Opportunities and Challenges. Diagnostics (Basel). 2023 Sep 26;13(19):3054. doi: 10.3390/diagnostics13193054. PMID 37835797
- [Background] Goyal H, Sherazi SAA, Gupta S, Perisetti A, Achebe I, Ali A, Tharian B, Thosani N, Sharma NR. Application of artificial intelligence in diagnosis of pancreatic malignancies by endoscopic ultrasound: a systemic review. Therap Adv Gastroenterol. 2022 Apr 29;15:17562848221093873. doi: 10.1177/17562848221093873. eCollection 2022. PMID 35509425